CLINICAL TRIAL: NCT05602740
Title: EPISODE-VS: hEad Pulse for Ischemic StrOke Verification Study
Brief Title: Detection of hEad Pulse for Ischemic StrOke Verification Study
Acronym: EPISODE_VS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: MindRhythm, Inc. (Industry)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor
Other Study IDs: EPISODE_VS
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-06

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MINDRHYTHM HARMONY: Passive Recording of the head pulse
  Interventions: Device: Harmony

INTERVENTIONS:
Device: Harmony — Passive recording of the head pulse

SUMMARY:
Prehospital providers encounter patients with suspected stroke frequently. Prehospital providers need tools to help triage large vessel stroke patients to comprehensive stroke centers. This device will identify large vessel stroke to ultimately improve triage decisions and optimize outcomes.

DETAILED DESCRIPTION:
Patients suspected of stroke by a prehospital provider will have a headset placed to record their headpulse during the encounter. These measurements will be used to assess the accuracy of the device at predicting the presence of large vessel occlusion (LVO) stroke. The MindRhythm, Inc., Harmony® 5000 device is intended to be used in the pre-hospital setting by medical professionals to diagnose large vessel occlusion stroke in adults suspected of having a stroke.

ELIGIBILITY:
Inclusion Criteria:

• suspected stroke in the prehospital setting

Exclusion Criteria:

* scalp laceration
* Patient refusal
* Prisoner, other vulnerable population
* Prehospital provider feels that the recording may interfere with care

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are being evaluated in the prehospital environment by Paramedics/EMTs in whom stroke is suspected.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
The primary effectiveness objective is to estimate the sensitivity and specificity of LVO diagnosis with Harmony®. | Through study completion, an average of 6 months
  The subject's final discharge diagnosis based on the CTA scan and the neurologist's assessment will serve as the "ground truth" diagnosis. The sensitivity and specificity will be estimated as the point estimate (Harmony® identified correctly divided by the ground truth number); the confidence intervals will be estimated by the Clopper-Pearson method (exact intervals for proportions).

CONTACTS AND LOCATIONS:
Overall Officials: James Paxton, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith WS, Keenan KJ, Lovoi PA. A Unique Signature of Cardiac-Induced Cranial Forces During Acute Large Vessel Stroke and Development of a Predictive Model. Neurocrit Care. 2020 Aug;33(1):58-63. doi: 10.1007/s12028-019-00845-x. PMID 31591693